CLINICAL TRIAL: NCT05795309
Title: Automated Insulin Delivery in Type 1 Diabetes Complicated by Gastroparesis
Acronym: AIDgastro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22HH8008
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Gastroparesis; Type 1 Diabetes
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Staggered randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid Automated Insulin Delivery (Experimental): The intervention is the Medtronic 780G Hybrid Automated Insulin Delivery system
  Interventions: Device: Hybrid Automated Insulin Delivery
- Standard care (No Intervention): The control is Standard Care with real-time CGM

INTERVENTIONS:
Device: Hybrid Automated Insulin Delivery — Consists of an insulin pump and real-time continuous glucose monitoring (CGM)
  Other Names: Medtronic 780G
  Arms: Hybrid Automated Insulin Delivery

SUMMARY:
This is a staggered randomised controlled trial that aims to assess the impact of an automated insulin delivery (AID) system on glucose, gastrointestinal and patient-reported outcomes.

DETAILED DESCRIPTION:
Following a run-in period of 2 weeks, participants will be randomised to control or hybrid automated insulin delivery (AID) using the 780G system and will remain in the intervention phase of the study for 12 weeks (4-week control, then 4-week AID or Control and finally 4-week AID). The total duration for each participant will be 14 weeks. There are 5 study visits (combination of face to face or/and remote) and two telephone visits in total.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years of age or older
* Type 1 diabetes confirmed on the basis of clinical features
* Type 1 diabetes for greater than 1 year
* On an intensified insulin regimen with multiple dose injection or insulin pump for > 3 months
* HbA1c >7.5% (58mmol/mol) (or %TIR 3.9-10mmol/L <52% for participants already using a continuous glucose sensor)
* Gastroparesis Cardinal Symptom Index (GCSI) ≥ 18 or evidence of delayed gastric emptying on nuclear medicine gastric emptying study

Exclusion Criteria:

* Enrolled in other clinical trials
* Estimated glomerular filtration rate of ≤30ml/min
* Pregnant or planning pregnancy
* Have active malignancy or under investigation for malignancy
* Severe visual impairment
* Reduced manual dexterity
* Use of any automated insulin delivery system
* Unable to participate due to other factors, as assessed by the Chief Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage time spent in glucose target (3.9-10mmol/L) | 4 - 8 weeks
  The change in percentage time in glucose target between baseline and intervention/control

SECONDARY OUTCOMES:
Percentage time spent in hypoglycaemia (<3.0mmol/L) | 4 - 8 weeks
  The change in percentage time in hypoglycaemia(<3.0mmol/L) between baseline and intervention/control
Percentage time spent in hypoglycaemia (<3.9mmol/L) | 4 - 8 weeks
  The change in percentage time in hypoglycaemia (<3.9mmol/L) between baseline and intervention/control
Percentage time spent in hyperglycaemia (>10mmol/L) | 4 - 8 weeks
  The change in percentage time in hyperglycaemia (>10mmol/L) between baseline and intervention/control

CONTACTS AND LOCATIONS:
Overall Officials: Nick Oliver, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London and Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No